CLINICAL TRIAL: NCT05300698
Title: MRI Versus Ocular UltraSonography for a Non Contact Evaluation of Ocular Layers
Acronym: MOUSE
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: YPL_2021_29
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Describe Ultrasound Matches and Disagreements Ocular and MRI
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — compare between MRI and ultrasound for indirect assessment of ocular layers
  Other Names: baseline

SUMMARY:
D0: inclusion visit

* information
* Realization of the ocular ultrasound (care)
* Collection of consent
* Realization of high resolution MRI with injection of contrast product (duration of 30 minutes) For the realization of the MRI, the contrast product used is the gadobutrol. The dose, the lowest allowing an enhancement of sufficient contrast for diagnostic purposes (0.1 mmol/kg body mass body), is administered as a bolus intravenously in the lying patient. The MRI examination can begin immediately after injection. The patient should be monitored for at least half an hour after this, the majority of undesirable effects occurring at the during this period. The indication of ocular ultrasound and ophthalmological follow-up of the patient up to 1 month after inclusion will be collected at from their medical records.

DETAILED DESCRIPTION:
D0: inclusion visit

* information
* Realization of the ocular ultrasound (care)
* Collection of consent
* Realization of high resolution MRI with injection of contrast product (duration of 30 minutes) For the realization of the MRI, the contrast product used is the gadobutrol. The dose, the lowest allowing an enhancement of sufficient contrast for diagnostic purposes (0.1 mmol/kg body mass body), is administered as a bolus intravenously in the lying patient. The MRI examination can begin immediately after injection. The patient should be monitored for at least half an hour after this, the majority of undesirable effects occurring at the during this period. The indication of ocular ultrasound and ophthalmological follow-up of the patient up to 1 month after inclusion will be collected at from their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Addressed in imaging for the realization of an ultrasound diagnostic eye
* Express consent to participate in the study
* Member of or beneficiary of a social security scheme

Exclusion Criteria:

* Patient with an absolute or relative contraindication to MRI (pacemaker or neurosensory stimulator or defibrillator implantable; ocular or cerebral ferromagnetic foreign body; claustrophobia)
* Absolute or relative contraindication to the injection of gadolinium (history of an allergic reaction to a product of contrast, bronchial asthma, allergic terrain, renal failure with serum creatinine clearance <30 mL/min)
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman: a pregnancy test in the woman of childbearing age is to be carried out before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited when they are referred for imaging to performing an ocular ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
description of concordance and discordance of ultrasound ocular and MRI | 1 DAY

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No